CLINICAL TRIAL: NCT04626726
Title: A Clinical Trial to Explore the Safety, Efficacy, and Remission Phase of CAR-T Cell in the Treatment of Adult Relapsed Refractory (R/R) Acute Lymphoblastic Leukemia Bridging Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Adult B-ALL Treated by CART Cell Bridging Allogeneic Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T for adult B-ALL
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Adult B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — fludarabine; fiu protein, E coli; Cyclophosphamide; Cholestanetriol 26-Monooxygenase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteers (Experimental): The patient voluntarily signs the informed consent, and the patient meets the entry criteria to diagnose patients with acute B lymphocytic leukemia expressing specific target antigens
  Interventions: Drug: CD19 CAR-T; Drug: CD22 CAR-T; Drug: CD19+CD22 CAR-T; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: CD19 CAR-T — CD19 CAR-T infusion for patients with CD19 positive tumor cells
  Other Names: Senl_19
Drug: CD22 CAR-T — CD22 CAR-T infusion for patients with CD22 positive tumor cells
  Other Names: Senl_22
Drug: CD19+CD22 CAR-T — CD19+CD22 CAR-T infusion for patients with CD19 positive and CD22 positive tumor cells
  Other Names: Senl_19+22
Drug: Fludarabine — 25mg/㎡ for D-4、D-3 and D-2
  Other Names: fiu
Drug: Cyclophosphamide — 500mg/㎡ for D-3 and D-2
  Other Names: ctx

SUMMARY:
This is an open, single-arm, phase I/phase II clinical study to evaluate efficacy and safety of chimeric antigen receptor T cell immunotherapy (CAR-T) in the treatment of Relapsed Refractory (R/R) adult acute lymphoblastic leukemia bridging allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
This trial openly recruited 50 patients into the group and were given CAR-T treatment. Patients participating in clinical trials will be tested and evaluated in terms of treatment safety, efficacy, and response duration. As assessed by clinicians, adult B-ALL patients who meet the enrollment criteria, after adequate communication, the patient or family members voluntarily join the clinical study, and are willing to bridge allogeneic hematopoiesis within 3 months after enrollment using CAR-T therapy。

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed a kind of Relapsed or Refractory Haematopoietic and Lymphoid Malignancies:
2. ECOG score≤2;
3. To be aged 1 to 65 years;
4. More than a month lifetime from the consent signing date.

Exclusion Criteria:

1. Serious cardiac insufficiency, left ventricular ejection fraction<50%;
2. Has a history of severe pulmonary function damaging;
3. Merging other progressing malignant tumor;
4. Merging uncontrolled infection;
5. Merging the metabolic diseases (except diabetes);
6. Merging severe autoimmune diseases or immunodeficiency disease;
7. Patients with active hepatitis B or hepatitis C;
8. Patients with HIV infection;
9. Has a history of serious allergies on Biological products (including antibiotics);
10. Has acute GvHD on allogeneic hematopoietic stem cell transplantation patients after stopping immunosuppressants a month;
11. Pregnancy or lactation women;
12. Any situation that would increase dangerousness of subjects or disturb the outcome of the clinical study according to the researcher's evaluation.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe/Adverse Events as a Measure of Safety | 28 days
  Number of Participants with Severe/Adverse Events as a Measure of Safety
Copies numbers of CAR in peripheral blood(PB) and/or bone marrow(BM) | 24 months
  Copies numbers of CAR in peripheral blood(PB) and/or bone marrow(BM)

SECONDARY OUTCOMES:
Objective response rate of complete remission and partial remission | 24 months
  Objective response rate of complete remission and partial remission
Overall survival time | 24 months
  Overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Luo, PhD&MD, Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- No.2 Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No